CLINICAL TRIAL: NCT06557499
Title: A Randomized, Data Analyst-masked, 3-way Cross-over, Pivotal Clinical Investigation to Evaluate the Performance of Two Polyurethane Male Condoms With Different Size and Thickness in Healthy Monogamous Couples During Vaginal Intercourse Compared With a Commercially Available Thin Latex Male Condom.
Brief Title: A 3-way Crossover Clinical Investigation to Assess the Performance of Two Different Sized Polyurethane Condoms Versus a Latex Condom in Healthy Monogamous Couples.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Reckitt Benckiser Healthcare (UK) Limited (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2628301
Record Dates: First submitted 2024-07-24; First posted 2024-08-16 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Contraception
Keywords: Condoms; Slippage; Breakage
MeSH Terms: interventions — Condoms

STUDY DESIGN:
Intervention Model Description: The condom types will be tested in a 3-way cross-over design where couples will be randomised to use each of the 3 condom types in a defined order, according to the randomisation schedule.
Who Masked: Outcomes Assessor
Masking Description: The clinical investigation is designed to be a data analyst-masked investigation where the data analyst who will perform the data analysis (both CRO and Sponsor staff involved in analysing the data) will not know which condom type couples have been randomised to use in each assessment period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Polyurethane (PU) male condom-Test condom 1 (Experimental)
  Interventions: Device: Polyurethane (PU) male condom-Test condom 1
- Polyurethane (PU) male condom-Test condom 2 (Experimental)
  Interventions: Device: Polyurethane (PU) male condom-Test condom 2
- Natural Rubber Latex (NRL) male condom- Control condom (Active Comparator)
  Interventions: Device: Natural Rubber Latex (NRL) male condom- Control condom

INTERVENTIONS:
Device: Polyurethane (PU) male condom-Test condom 1 — A minimum of 5 condoms (maximum 7 condoms) of each condom type will be provided to couples to be used during vaginal intercourse over a maximum 5-week period (assessment period). Couples will repeat the assessment period for each of the 3 condom types.
  Arms: Polyurethane (PU) male condom-Test condom 1
Device: Polyurethane (PU) male condom-Test condom 2 — A minimum of 5 condoms (maximum 7 condoms) of each condom type will be provided to couples to be used during vaginal intercourse over a maximum 5-week period (assessment period). Couples will repeat the assessment period for each of the 3 condom types.
  Arms: Polyurethane (PU) male condom-Test condom 2
Device: Natural Rubber Latex (NRL) male condom- Control condom — A minimum of 5 condoms (maximum 7 condoms) of each condom type will be provided to couples to be used during vaginal intercourse over a maximum 5-week period (assessment period). Couples will repeat the assessment period for each of the 3 condom types.
  Arms: Natural Rubber Latex (NRL) male condom- Control condom

SUMMARY:
This investigation is designed to evaluate the performance rate of two polyurethane male condoms with different sizes and thicknesses versus a standard natural rubber latex (NRL) male condom.

The purpose of this study is to see how well the experimental condoms perform compared to the latex rubber condom (for example, how often the different condom types break or slip off the penis).

Sponsor also wants to find out how well couples like using the three condom types and whether they experience any problems when using the condoms (for example, irritation or discomfort).

DETAILED DESCRIPTION:
In this clinical investigation, new two PU male condoms (test condoms) will be evaluated against a marketed NRL male condom (control condom). This clinical investigation will also evaluate the in-use tolerance of the test and control condoms.

ELIGIBILITY:
Inclusion Criteria:

1. Both partners participating must provide written informed consent.
2. Couples must include a male and female within a heterosexual couple and be between 18 - 60 years of age inclusive.
3. Both partners must be willing to respond to questions about their reproductive and contraceptive history and use of condoms during interviews and respond to self-administered questionnaires as per instructions.
4. Both partners must agree to answer the questions in the condom use questionnaires and two scales as soon as possible and within 2 (+6) hours following each coital act.
5. Both partners must be generally healthy and in a mutually monogamous heterosexual relationship - current relationship ≥ 3 months.
6. All couples must be averaging one act of intercourse weekly, agree to have penile-vaginal intercourse with a frequency sufficient to meet CIP requirements (a minimum of 5 coital acts over 5 weeks per assessment period-).
7. The female partner must also use an established (as agreed by the Investigator) other highly effective form of non-barrier contraception, unless post-menopausal (confirmed menopausal prior to screening, amenorrhea for at least 12 months after cessation of exogenous hormone treatment) in which case no second form of contraception is required. Highly effective non-barrier contraception includes oral contraceptive (oestrogen and progestogen or progestogen-only hormonal contraception associated with inhibition of ovulation), intra-uterine device (IUD) or intra-uterine system (IUS), hormonal implant, injectables, patch and or sterilization of at least one partner (i.e., bilateral tubal ligation, vasectomy deemed medically successful).
8. Both partners must be able to understand instructions for correct use of condoms.
9. Both partners must have an adequate level of literacy to understand and to be able to answer the questionnaires.
10. Both partners must agree to use only the investigational condoms during the time of participation.
11. Participants must agree to use the penis measuring kit provided to measure the erect penis at investigation start.
12. Both partners must agree not to use drugs or non-investigational devices that can affect sexual performance.
13. Both partners must have no known sexually transmitted infections including Human Immunodeficiency Virus (HIV) / acquired immune deficiency syndrome (AIDS) (medical history via self-report) (uncomplicated Herpes simplex virus (HSV) and positive Human papillomavirus (HPV) which areis asymptomatic may be included in the investigation study in the opinion of the Investigator).
14. Both partners must agree to use only lubricant(s) provided for the duration of investigation.
15. Both partners must agree not to wear any genital piercing jewellery for the duration of the clinical investigation.
16. Both partners must have no past medical history of any health condition (self-reported) that, in the opinion of the Investigator, would be considered clinically relevant.
17. Couples must have a compatible electronic device with internet access which they are willing to upload questionnaire data to the web-based platform throughout the investigation.
18. Both partners will be available for follow-up.

Exclusion Criteria:

1. Either partner is or becomes aware of an allergy or sensitivity to the ingredients of any of the products, including the test or control condoms or any lubrication products provided.
2. Either partner has been receiving daily treatment for their pre-existing skin condition (for example, severe eczema/psoriasis) within the three months prior to the screening for this study.
3. Female partner that is pregnant or desires to become so while participating in investigation, (females of childbearing potential must have a negative pregnancy test as part of screening).
4. Any couple undergoing any form of fertility treatment such as in-vitro fertilisation.
5. Either partner needs to use condoms for sexually transmitted infection (STI) protection (e.g., discordance for Human Immunodeficiency Virus (HIV) or herpes).
6. Either partner has previous or planned genital surgery that in the opinion of the Investigator would consider the participant unsuitable to participate in the clinical investigation (e.g., laser for abnormal smear).
7. Either partner are commercial sex workers.
8. Either partner are itinerant persons who will be unable to complete the clinical investigation (e.g., migrant farm workers).
9. Couples that in the opinion of the Investigator, would be unable to complete the investigation.
10. Male partners that have known erectile or ejaculatory dysfunction in the past month.
11. Either partner requires to use/ is using medication or preparations that are applied topically to the genitalia area or intravaginally, other than that supplied for the investigation.
12. A female partner that has been diagnosed with or treated for vaginal complaints (including vaginal dryness) in the previous 3 months which, in the opinion of the Investigator, deems the partner unsuitable for the investigation.
13. Either partner uses any medication which in the investigator's opinion may interfere with the use of condoms.
14. A male partner with abnormal penile anatomy or genital lesion (e.g., balanoposthitis) that would, in the opinion of the Investigator, affect the ability to keep the condom in place during intercourse.
15. Either partner is suffering from any health conditions (self-reported) or any condition which could, in the opinion of the Investigator, affect the outcome of the investigation or affect their safety if they participate.
16. Either partner have participated in a clinical trial in the previous month which could, in the opinion of the Investigator, affect the outcome of the investigation.
17. Either partner is an employee of the investigational Sponsor or affiliated with the clinical research centre (i.e., enrolment of the Investigator, his/ her family members, employees and other dependent persons).
18. Either partner has a recent history of drug/alcohol abuse within the previous 12 months.
19. Either partner has an inability to follow the procedures of the investigation, (e.g., due to language problems, psychological disorders, health conditions such as dementia).
20. Either partner is unable, in the opinion of the Investigator, to fully comply with the investigation requirements.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 600 (Estimated)
Dates: Start 2024-08-23 (Actual); Primary Completion 2025-05-19 (Estimated); Study Completion 2025-05-19 (Estimated)

PRIMARY OUTCOMES:
Total clinical failure rate of Polyurethane (PU) male (Test condom 1) condom compared to Natural Rubber Latex (NRL) male condom. | within 8 hours following each coital act for each condom use
  The total clinical failure rate (combined breakage and slippage) of PU male test condom (Test condom 1) compared to the NRL male control condom.
  Clinical failure rate is calculated as the number of condoms with at least 1 acute clinical failure event divided by the number of condoms used during intercourse, reported as a percentage. Clinical failure events, defined in ISO 29943-1:2017, will be reported by participants.
Total clinical failure rate of Polyurethane (PU) male (Test condom 2) condom compared to Natural Rubber Latex (NRL) male condom. | within 8 hours following each coital act for each condom use
  The total clinical failure rate (combined breakage and slippage) of PU male test condom (Test condom 2) compared to the NRL male control condom.
  Clinical failure rate is calculated as the number of condoms with at least 1 acute clinical failure event divided by the number of condoms used during intercourse, reported as a percentage. Clinical failure events, defined in ISO 29943-1:2017, will be reported by participants.

SECONDARY OUTCOMES:
Clinical breakage rate of PU Male Test Condom 1 compared to NRL male control condom | within 8 hours following each coital act for each condom use
  The total clinical breakage rate of the PU male test condom (Test condom 1) compared to the NRL male control condom when used during vaginal intercourse.
  The total clinical breakage rate is determined from the number of condoms broken or torn during vaginal intercourse or withdrawal from the vagina divided by the number of condoms used during intercourse, reported as a percentage.
Clinical slippage rate of PU Male Test Condom 1 compared to NRL male control condom | within 8 hours following each coital act for each condom use
  The total clinical slippage rate of the PU male test condom (Test condom 1) compared to the NRL male control condom when used during vaginal intercourse.
  The total clinical slippage rate is determined from the number of condoms that slipped completely off the penis during intercourse or withdrawal from the vagina, divided by the number of condoms used during vaginal intercourse, reported as a percentage.
Clinical breakage rate of PU Male Test Condom 2 compared to NRL male control condom | within 8 hours following each coital act for each condom use
  The total clinical breakage rate of the PU male test condom (Test condom 2) compared to the NRL male control condom when used during vaginal intercourse.
  The total clinical breakage rate is determined from the number of condoms broken or torn during vaginal intercourse or withdrawal from the vagina divided by the number of condoms used during intercourse, reported as a percentage.
Clinical slippage rate of PU Male Test Condom 2 compared to NRL male control condom | within 8 hours following each coital act for each condom use
  The total clinical slippage rate of the PU male test condom (Test condom 2) compared to the NRL male control condom when used during vaginal intercourse.
  The total clinical slippage rate is determined from the number of condoms that slipped completely off the penis during intercourse or withdrawal from the vagina, divided by the number of condoms used during vaginal intercourse, reported as a percentage.
Non-clinical breakage rate for each of the PU male condoms (test condom 1 and test condom 2) and the NRL male control condom. | within 8 hours following each coital act for each condom use
  The total non-clinical breakage rate for each of the PU male test condom and the NRL male control condom when used during vaginal intercourse.
  The total non-clinical breakage rate is determined from the number of condoms that tear during handling.
Non-clinical slippage respectively of each PU male test condom (test condom 1 and test condom 2) and the NRL male control condom. | within 8 hours following each coital act for each condom use
  The total non-clinical slippage rate for each of the PU male test condoms and the NRL male control condom when used during vaginal intercourse.
  The total non-clinical slippage rate is determined from the number of observations where the user fails to hold onto the condom at the base of the penis during withdrawal and/ or because the user delayed withdrawal after sex.
User acceptability of the 2 PU male test condoms (test condom 1 and test condom 2) and the NRL male control condom. | within 8 hours following each coital act for each condom use
  User acceptability, experience, and preference for each condom type will be evaluated through participant-perceived questions.
  Participant's experience on the use of each type of condoms [Acceptability as assessed by participant perceived questionnaires (designed by following ISO 29943-1)
In-use tolerability of the 2 PU male test condoms (test condom 1 and test condom 2) and the NRL male control condom. | 5 weeks for each condom type
  The in-use tolerability of each condom type will be evaluated through participant-perceived questions (designed by following ISO 29943-1).

CONTACTS AND LOCATIONS:
Overall Officials: Terri Walsh, Principal Investigator — Essential Access Health
Locations (3):
- United States (3):
  - Essential Access Health-Berkeley, Berkeley, California
  - Essential Access Health -Los Angeles, Los Angeles, California
  - Essential Acess Health- Seattle, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No